CLINICAL TRIAL: NCT05234021
Title: HER2-directed Biosimilar OgivriTM in Breast Cancer: Real World Observational Trial for the Description of Quality of Life and Outcome Using ePRO (OGIPRO- Trial)
Brief Title: HER2-directed Biosimilar in Breast Cancer: Real World ePRO
Acronym: OGIPRO
Status: Completed | Type: Observational
Sponsor: OnkoZentrum Zürich AG (Other)
Collaborators: University of Zurich (Other); Palleos Healthcare GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: KEK 2021-D0051
Record Dates: First submitted 2022-01-04; First posted 2022-02-10 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: HER2-positive Breast Cancer; Biosimilar; Patient Reported Outcome
Keywords: ePRO; HER2; Breast Cancer; Biosimilar; Patient Reported Outcome; APP
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project will engage anti-HER2 directed Trastuzumab biosimilar with a novel quality of ePRO and enable comparison of reliable reference real world patient data, thereby creating a basis for analytic research in order to promote the quality and efficiency of treatment

DETAILED DESCRIPTION:
Comprehensive data on patient history and follow-up modalities, AEs and outcome will be collected as ePRO to provide high-quality reports and quantitatively abundant data provided by patients. In particular, prospectively collected data shall be compared to previously collected ePRO from women treated for HER2-positive BC in a variety of indications and settings . Since a large number of data entries for wellbeing and symptom reporting (according to CTCAE) is available from these patients, the investigators will refer to this as a historic registry data warehouse. Accordingly, the ePRO from these patients treated for HER2 positive BC are available for planned comparative analysis and shall be applied to indicate differences in anti-HER2 directed medication between Ogivri and Herceptin.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Patients ≥ 18 years
* Patients with HER2-positive breast cancer (IHC-FISH/SISH)
* Undergoing Anti-HER2 treatment during the observational period containing OgivriTM (Trastuzumab) +/- Pertuzumab +/- Chemotherapy
* Personal smartphone with iOS or Android system. The operating system must be updated to one of the two newest main versions

Exclusion Criteria:

* Patients, whose compliance to the studies' protocol, e.g. due to mental health problems, physical problems, or the private life situation, can be justifiably doubted
* Patients with insufficient knowledge about the use of a smartphone

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: HER2 positive Breast cancer patients undergoing Anti-HER2 treatment with Ogivri
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Number of adverse events (AE) according to the Common Terminology Criteria for Adverse Events (CTCAE) | six weeks
  AEs according to the Common Terminology Criteria for Adverse Events (CTCAE) after six weeks as documented by the patients as ePRO via Consilium CareTM app.
Severity of adverse events (AE) according to the Common Terminology Criteria for Adverse Events (CTCAE) | six weeks
  AEs according to the Common Terminology Criteria for Adverse Events (CTCAE) after six weeks as documented by the patients as ePRO via Consilium CareTM app.

SECONDARY OUTCOMES:
Wellbeing | six weeks
  According to grades 0-4 (avoiding grade 5 = death) of an ECOG (Eastern Cooperative Oncology Group) Performance Status Scale, here the values are: min 0.1; max 10: higher scores in the particular utility arrangement on this app mean a better outcome.
EQ-5D-5L (European Quality of Life 5 Dimensions 5 Level Version); descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain and anxiety. Each dimension has 5 levels: (min 1; max 5); higher scores mean a worse outcome. | six weeks
  Quality of Live questionnaire will be sent to patients q 3 weeks
Unplanned Consultations | nine weeks
  Unplanned consultations are defined as additional consultations outside of planned therapy or control visits

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Trojan, M.D., Principal Investigator — Seespital Horgen
Locations (3):
- Switzerland (3):
  - Andreas Trojan, Horgen, Canton of Zurich
  - ZeTup, Rapperswil-Jona
  - Onkologiepraxis Bellvue, Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Trojan A, Roth S, Atassi Z, Kiessling M, Zenhaeusern R, Kadvany Y, Schumacher J, Kullak-Ublick GA, Aapro M, Eniu A. Comparison of the Real-World Reporting of Symptoms and Well-Being for the HER2-Directed Trastuzumab Biosimilar Ogivri With Registry Data for Herceptin in the Treatment of Breast Cancer: Prospective Observational Study (OGIPRO) of Electronic Patient-Reported Outcomes. JMIR Cancer. 2024 Apr 4;10:e54178. doi: 10.2196/54178. PMID 38573759